CLINICAL TRIAL: NCT07260903
Title: Can Photobiomodulation Improve Balance and Cognition in Individuals Over 60: a Pilot Feasibility Placebo Randomized Controlled Trial.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Central Lancashire (Other)
Responsible Party: Principal Investigator, Jonathan Sinclair, Professor, University of Central Lancashire
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PMB balance and cognition
Record Dates: First submitted 2025-11-21; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Age >60
MeSH Terms: interventions — Low-Level Light Therapy; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham photobiomodulation (Sham Comparator): 8-weeks sham photobiomodulation.
  The sham device will follow the same protocol but without active light emission.
  Interventions: Other: Sham 8-weeks photobiomodulation
- Photobiomodulation (Experimental): 8-weeks photobiomodulation
  Twenty-four-minute photobiomodulation stimulation (twelve minutes at 670 nm followed by twelve minutes at 810 nm). Three times per week for 8-weeks.
  Interventions: Device: Photobiomodulation

INTERVENTIONS:
Device: Photobiomodulation — 8-weeks photobiomodulation
  Arms: Photobiomodulation
Other: Sham 8-weeks photobiomodulation — The sham device will follow the same protocol but without active light emission.
  Arms: Sham photobiomodulation

SUMMARY:
As people age, changes in balance and memory can make daily life more difficult and increase the risk of falls. Falls are one of the main causes of injury, hospitalization and loss of independence in older adults, while even mild declines in memory and concentration can reduce confidence, social participation and overall quality of life. Therefore, safe, affordable, and practical ways to help older adults remain steady on their feet and mentally sharp are urgently needed.

The aim of this project is therefore to conduct a pilot feasibility randomized controlled trial to examine whether regular home-based photobiomodulation can improve balance and cognitive function in adults aged over 60. If successful, this research could help shape future strategies for preventing falls, enhancing wellbeing and maintaining independence in older people.

ELIGIBILITY:
Inclusion Criteria:

* Aged from 60-80 years
* Ability to complete written questionnaires independently
* Able to provide informed consent

Exclusion Criteria:

* Current or past history of head injury
* Use of medications acting on the central nervous system
* Active skin conditions on the forehead or scalp
* Ongoing brain stimulation therapy
* History of migraines
* Sensitive skin, allergies

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-07-10 (Estimated)

PRIMARY OUTCOMES:
n-1-back (deviation) | Baseline
  The n-1-back (deviation) task is a working memory test where participants respond when the current stimulus differs from the one presented n-1 trials earlier.
n-1-back (deviation) | 1 hour
  The n-1-back (deviation) task is a working memory test where participants respond when the current stimulus differs from the one presented n-1 trials earlier.
n-1-back (deviation) | 8-weeks
  The n-1-back (deviation) task is a working memory test where participants respond when the current stimulus differs from the one presented n-1 trials earlier.

SECONDARY OUTCOMES:
n-2-back (deviation) | Baseline
  The n-2-back (deviation) task is a working memory test where participants respond when the current stimulus differs from the one presented n-2 trials earlier.
n-2-back (deviation) | 1 hour
  The n-2-back (deviation) task is a working memory test where participants respond when the current stimulus differs from the one presented n-2 trials earlier.
n-2-back (deviation) | 8-weeks
  The n-2-back (deviation) task is a working memory test where participants respond when the current stimulus differs from the one presented n-2 trials earlier.
n-1-back (post-deviation) | Baseline
  The n-1-back (post-deviation) task assesses working memory performance on the trial immediately following a deviation from the stimulus presented n-1 trials earlier.
n-1-back (post-deviation) | 1 hour
  The n-1-back (post-deviation) task assesses working memory performance on the trial immediately following a deviation from the stimulus presented n-1 trials earlier.
n-1-back (post-deviation) | 8-weeks
  The n-1-back (post-deviation) task assesses working memory performance on the trial immediately following a deviation from the stimulus presented n-1 trials earlier.
n-2-back (post-deviation) | Baseline
  The n-2-back (post-deviation) task assesses working memory performance on the trial immediately following a deviation from the stimulus presented n-2 trials earlier.
n-2-back (post-deviation) | 1 hour
  The n-2-back (post-deviation) task assesses working memory performance on the trial immediately following a deviation from the stimulus presented n-2 trials earlier.
n-2-back (post-deviation) | 8-weeks
  The n-2-back (post-deviation) task assesses working memory performance on the trial immediately following a deviation from the stimulus presented n-2 trials earlier.
n-1-back (post-target) | Baseline
  The n-1-back (post-target) task assesses working memory performance on the trial immediately following a target that matched the stimulus presented n-1 trials earlier.
n-1-back (post-target) | 1 hour
  The n-1-back (post-target) task assesses working memory performance on the trial immediately following a target that matched the stimulus presented n-1 trials earlier.
n-1-back (post-target) | 8-weeks
  The n-1-back (post-target) task assesses working memory performance on the trial immediately following a target that matched the stimulus presented n-1 trials earlier.
n-2-back (post-target) | Baseline
  he n-2-back (post-target) task assesses working memory performance on the trial immediately following a target that matched the stimulus presented n-2 trials earlier.
n-2-back (post-target) | 1 hour
  he n-2-back (post-target) task assesses working memory performance on the trial immediately following a target that matched the stimulus presented n-2 trials earlier.
n-2-back (post-target) | 8-weeks
  he n-2-back (post-target) task assesses working memory performance on the trial immediately following a target that matched the stimulus presented n-2 trials earlier.
n-1-back (load) | Baseline
  The n-1-back (load) condition measures working memory performance under the cognitive demand of tracking stimuli 1 trial back.
n-1-back (load) | 1 hour
  The n-1-back (load) condition measures working memory performance under the cognitive demand of tracking stimuli 1 trial back.
n-1-back (load) | 8-weeks
  The n-1-back (load) condition measures working memory performance under the cognitive demand of tracking stimuli 1 trial back.
n-2-back (post-load) | Baseline
  The n-2-back (post-load) condition assesses working memory performance on the trial immediately following a high cognitive load in the n-2-back task.
n-2-back (post-load) | 1 hour
  The n-2-back (post-load) condition assesses working memory performance on the trial immediately following a high cognitive load in the n-2-back task.
n-2-back (post-load) | 8-weeks
  The n-2-back (post-load) condition assesses working memory performance on the trial immediately following a high cognitive load in the n-2-back task.
Coop-Wonka chart | Baseline
  The Coop-Wonka chart is a six item questionnaire with a 1-5 scoring system for each thus the chart has a maximum score of 30 which indicates the lowest possible psychological Wellbeing.
Coop-Wonka chart | 1 hour
  The Coop-Wonka chart is a six item questionnaire with a 1-5 scoring system for each thus the chart has a maximum score of 30 which indicates the lowest possible psychological Wellbeing.
Coop-Wonka chart | 8-weeks
  The Coop-Wonka chart is a six item questionnaire with a 1-5 scoring system for each thus the chart has a maximum score of 30 which indicates the lowest possible psychological Wellbeing.
Beck Depression Inventory | Baseline
  Psychological wellbeing - the Beck Depression Inventory is a 21 questionnaire with questions that range in scoring from 0-3, thus the maximum score is 63 which is the highest depression score possible.
Beck Depression Inventory | 1 hour
  Psychological wellbeing - the Beck Depression Inventory is a 21 questionnaire with questions that range in scoring from 0-3, thus the maximum score is 63 which is the highest depression score possible.
Beck Depression Inventory | 8-weeks
  Psychological wellbeing - the Beck Depression Inventory is a 21 questionnaire with questions that range in scoring from 0-3, thus the maximum score is 63 which is the highest depression score possible.
Pittsburgh Sleep Quality Index | Baseline
  The Pittsburgh Sleep Quality index, is a questionnaire that consists of 19 self-rated questions, grouped into 7 components. Each component is scored separately, weighted equally on a 0 - 3 scale and the scores of the 7 components are then added to give a global score, which has a range of 0 - 21 with higher scores indicating worse sleep quality.
Pittsburgh Sleep Quality Index | 1 hour
  The Pittsburgh Sleep Quality index, is a questionnaire that consists of 19 self-rated questions, grouped into 7 components. Each component is scored separately, weighted equally on a 0 - 3 scale and the scores of the 7 components are then added to give a global score, which has a range of 0 - 21 with higher scores indicating worse sleep quality.
Pittsburgh Sleep Quality Index | 8-weeks
  The Pittsburgh Sleep Quality index, is a questionnaire that consists of 19 self-rated questions, grouped into 7 components. Each component is scored separately, weighted equally on a 0 - 3 scale and the scores of the 7 components are then added to give a global score, which has a range of 0 - 21 with higher scores indicating worse sleep quality.
State Trait Anxiety Inventory | Baseline
  The state trait anxiety inventory is a 40 item questionnaire with each question having a 1-4 score system, thus the maximum score is 80 which indicates the highest level of anxiety.
State Trait Anxiety Inventory | 1 hour
  The state trait anxiety inventory is a 40 item questionnaire with each question having a 1-4 score system, thus the maximum score is 80 which indicates the highest level of anxiety.
State Trait Anxiety Inventory | 8-weeks
  The state trait anxiety inventory is a 40 item questionnaire with each question having a 1-4 score system, thus the maximum score is 80 which indicates the highest level of anxiety.
Insomnia Severity Index | Baseline
  The Insomnia Severity Index is a brief instrument designed to assess the severity of both nighttime and daytime components of insomnia. The Insomnia Severity Index is a 7-item self-report questionnaire yielding a total score ranging from 0 to 28.
Insomnia Severity Index | 1 hour
  The Insomnia Severity Index is a brief instrument designed to assess the severity of both nighttime and daytime components of insomnia. The Insomnia Severity Index is a 7-item self-report questionnaire yielding a total score ranging from 0 to 28.
Insomnia Severity Index | 8-weeks
  The Insomnia Severity Index is a brief instrument designed to assess the severity of both nighttime and daytime components of insomnia. The Insomnia Severity Index is a 7-item self-report questionnaire yielding a total score ranging from 0 to 28.
Epworth Sleepiness Scale | Baseline
  The Epworth Sleepiness Scale is a self-administered questionnaire with 8 questions. Respondents are asked to rate, on a 4-point scale (0-3) with a maximum score of 24.
Epworth Sleepiness Scale | 1 hour
  The Epworth Sleepiness Scale is a self-administered questionnaire with 8 questions. Respondents are asked to rate, on a 4-point scale (0-3) with a maximum score of 24.
Epworth Sleepiness Scale | 8-weeks
  The Epworth Sleepiness Scale is a self-administered questionnaire with 8 questions. Respondents are asked to rate, on a 4-point scale (0-3) with a maximum score of 24.
Everyday Memory Errors Questionnaire | Baseline
  The Everyday Memory Errors Questionnaire is a brief self-report instrument designed to assess the frequency of memory lapses in daily life. It consists of multiple items that yield a total score reflecting the extent of everyday memory difficulties.
Everyday Memory Errors Questionnaire | 1 hour
  The Everyday Memory Errors Questionnaire is a brief self-report instrument designed to assess the frequency of memory lapses in daily life. It consists of multiple items that yield a total score reflecting the extent of everyday memory difficulties.
Everyday Memory Errors Questionnaire | 8-weeks
  The Everyday Memory Errors Questionnaire is a brief self-report instrument designed to assess the frequency of memory lapses in daily life. It consists of multiple items that yield a total score reflecting the extent of everyday memory difficulties.
Falls Efficacy | Baseline
  The Falls Efficacy Scale is a brief self-report instrument designed to assess confidence in performing daily activities without falling. It consists of multiple items that yield a total score reflecting fear of falling and perceived fall-related self-efficacy.
Falls Efficacy | 1 hour
  The Falls Efficacy Scale is a brief self-report instrument designed to assess confidence in performing daily activities without falling. It consists of multiple items that yield a total score reflecting fear of falling and perceived fall-related self-efficacy.
Falls Efficacy | 8-weeks
  The Falls Efficacy Scale is a brief self-report instrument designed to assess confidence in performing daily activities without falling. It consists of multiple items that yield a total score reflecting fear of falling and perceived fall-related self-efficacy.
Anterior-posterior balance | Baseline
  The maximum anterior-posterior displacement of the centre of pressure during a two-minute balance task.
Anterior-posterior balance | 1 hour
  The maximum anterior-posterior displacement of the centre of pressure during a two-minute balance task.
Anterior-posterior balance | 8-weeks
  The maximum anterior-posterior displacement of the centre of pressure during a two-minute balance task.
Medio-lateral balance | Baseline
  The maximum medio-lateral displacement of the centre of pressure during a two-minute balance task.
Medio-lateral balance | 1 hour
  The maximum medio-lateral displacement of the centre of pressure during a two-minute balance task.
Medio-lateral balance | 8-weeks
  The maximum medio-lateral displacement of the centre of pressure during a two-minute balance task.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Central Lancashire, Preston, Lancashire, United Kingdom

IPD SHARING:
Plan to Share IPD: No